CLINICAL TRIAL: NCT02106000
Title: An Enabling Study to Compare the Inhalation Profiles of Women in the Third Stage of Labour to Those of Non-pregnant Female Volunteers and to Explore Whether There Are Any Differences Which Could Impact the Delivery of an Inhaled Medicinal Product
Brief Title: A Non-investigational Product (IP) Study to Investigate Lung Function in Women in the Third Stage of Labour
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201248
Record Dates: First submitted 2014-04-03; First posted 2014-04-07 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Haemorrhage
Keywords: Post Partum; Inhaled Oxytocin; Inhalation Profiles
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm 1: Non-pregnant females: Inhalation profiles will be recorded for non-pregnant females
  Interventions: Device: Inhalation profile recorder
- Arm 2: Pregnant females: Inhalation profiles will be recorded for the women in the 3rd stage of labour
  Interventions: Device: Inhalation profile recorder

INTERVENTIONS:
Device: Inhalation profile recorder — Up to three inhalation profiles will be recorded whilst inhaling with maximal effort

SUMMARY:
The purpose of this study is to record and compare the inhalation profiles of non pregnant women and those who are in the third stage of labour. The inhalation profiles will be recorded from consenting women as they inhale with maximal effort through an inhalation profile recorder [Glaxosmithkline (GSK), Ware]. The recorder will simulate resistance to airflow and will be representative of a dry powder inhaler of moderate resistivity. The inhalation endpoints will include Peak Pressure Drop, Peak Inspiratory Flow Rate, Inhaled Volume, Inhalation time, Average Inhalation Flow Rate and Acceleration rate which will be compared between the two female cohorts. Inhalation profiles recorded in this way may subsequently be used to study the in-vitro performance of investigational materials across inhalation parameters representative of the target patient population.

An appropriate number of subjects will be consented so that approximately 40 subjects (20 non-pregnant females and 20 stage three labour subjects) complete assessments. The inhalation profiles will be recorded on the same day of screening or at another time within a span of 50 days

ELIGIBILITY:
Inclusion Criteria:

* A non-pregnant female subject is eligible to participate in the study if she is in the age group of 18 to 30 years (inclusive), at the time of signing the informed consent; is healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history; is having a body weight >= 50 kilogram (kg) and Body Mass Index (BMI) within the range 19 - 29.9 kg/meter^2 (inclusive); is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form; OR is having a clinical abnormality which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GSK Medical Monitor, if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Pregnant Female will be eligible to participate in the study if she belongs to the age group of 18 to 30 years (inclusive), at the time of signing the informed consent; is healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history; is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form ;OR is having a clinical abnormality which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GSK Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.

Exclusion Criteria:

* Healthy Volunteers will be excluded from the study if they have a history or regular use of tobacco or smoking products within 6 months prior to screening; have a current history of Asthma or history of lung disease; have a history of Airway obstruction or abnormality OR have an upper or lower respiratory tract infection within four weeks of the inhalation assessment visit.
* Pregnant Females will be excluded from the study if they are undergoing Caesarean Section; OR have preeclampsia; have an upper or lower respiratory tract infection within four weeks of the inhalation assessment visit; are receiving an epidural or opioid analgesia for pain management; OR require instrumental or otherwise assisted delivery as assessed by the midwife staff at time of inhalation assessment visit OR have a current history of asthma or lung disease ; have a history of airway obstruction or abnormality; OR have a history or regular use of tobacco or smoking products within 6 months prior to screening

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women: pregnant and non-pregnant non-pregnant female subject is eligible to participate in the study if she is in the age group of 18 to 30 years pregnant female will be eligible to participate in the study if she belongs to the age group of 18 to 30 years
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2014-12-20 (Actual); Study Completion 2014-12-20 (Actual)

PRIMARY OUTCOMES:
Characterization of the inhalation profile of non-pregnant women by measuring Peak pressure drop | Screening, Up to Day 50
  Up to three inhalation profiles will be recorded in the semi-supine position and the assessment will be carried out by measuring the Peak pressure Drop (kPa) using the inhalation profile recorder
Characterization of the inhalation profile of non-pregnant women by measuring Peak Inspiratory Flow Rate | Screening, Up to Day 50
  Up to three inhalation profiles will be recorded in the semi-supine position and the assessment will be carried out for Peak Inspiratory Flow Rate [Liters/minute (L/min)] using the inhalation profile recorder
Characterization of the inhalation profile of non-pregnant women by measuring Inhaled Volume | Screening, Up to Day 50
  Up to three inhalation profiles will be recorded in the semi-supine position and the assessment will be carried out for the Inhaled Volume (L) using the inhalation profile recorder
Characterization of the inhalation profile of non-pregnant women by measuring Inhalation time | Screening, Up to Day 50
  Up to three inhalation profiles will be recorded in the semi-supine position and the assessment will be carried out for the Inhalation time measured in seconds(s)
Characterization of the inhalation profile of non-pregnant women by measuring Average Inhalation Flow Rate | Screening, Up to Day 50
  Up to three inhalation profiles will be recorded in the semi-supine position and the assessment will be carried out for Average Inhalation Flow Rate (L/min) measured using the inhalation profile recorder
Characterization of the inhalation profile of non-pregnant women by measuring Acceleration rate | Screening, Up to Day 50
  Up to three inhalation profiles will be recorded in the semi-supine position and the assessment of Acceleration rate (L/min/s) will be measured using the inhalation profile recorder
Characterization of the inhalation profile of women in the 3rd stage of labour by measuring Peak pressure Drop | Screening, Up to Day 50
  Up to three inhalation profiles will be recorded in a comfortable position (the position will be recorded) and the assessment will be carried out by measuring the Peak pressure Drop (kPa) using the inhalation profile recorder
Characterization of the inhalation profile of women in the 3rd stage of labour by measuring Peak Inspiratory Flow Rate | Screening, Up to Day 50
  Up to three inhalation profiles will be recorded in a comfortable position (the position will be recorded) and the assessment will be carried out for Peak Inspiratory Flow Rate (L/min) using the inhalation profile recorder
Characterization of the inhalation profile of women in the 3rd stage of labour by measuring Inhaled Volume | Screening, Up to Day 50
  Up to three inhalation profiles will be recorded in a comfortable position (the position will be recorded) and the assessment will be carried out for the Inhaled Volume (L) using the inhalation profile recorder
Characterization of the inhalation profile of women in the 3rd stage of labour by measuring Inhalation time | Screening, Up to Day 50
  Up to three inhalation profiles will be recorded in a comfortable position (the position will be recorded) and the assessment will be carried out for the Inhalation time measured in seconds
Characterization of the inhalation profile of women in the 3rd stage of labour by measuring Average Inhalation Flow Rate | Screening, Up to Day 50
  Up to three inhalation profiles will be recorded in a comfortable position (the position will be recorded) and the assessment will be carried out for Average Inhalation Flow Rate (L/min) measured using the inhalation profile recorder
Characterization of the inhalation profile of women in the 3rd stage of labour by measuring Acceleration rate | Screening, Up to Day 50
  Up to three inhalation profiles will be recorded in a comfortable position (the position will be recorded) and the assessment of Acceleration rate (L/min/s) will be measured using the inhalation profile recorder

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- See also: Results for study 201248 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201248?search=study&search_terms=201248#rs